CLINICAL TRIAL: NCT01076517
Title: A Humanitarian Device Exemption Treatment Protocol of TheraSphere For Treatment of Unresectable Hepatocellular Carcinoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Stanford University (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Daniel Yung-Ho Sze, Professor of Radiology, Stanford University
Other Study IDs: IRB-14324 (NOT RESEARCH); HEP0016 (Other: OnCore)
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

INTERVENTIONS:
Device: Therasphere — Beta-emitting 90yttrium encapsulated in glass microspheres for intraarterial administration to the liver.
  Other Names: HCC; hepatocellular carcinoma treatment

SUMMARY:
To provide Therasphere treatment for patients diagnosed with unresectable liver cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients of any age, of any race or sex, who have hepatocellular carcinoma of the liver, and who are able to give informed consent, will be eligible. Patients must have an ECOG Performance Status score of </= 2, with a life expectancy of >/= 3 months, non-pregnant with an acceptable contraception in premenopausal women. Patients must be >4 weeks since prior radiation or prior surgery and at least 1 month post other chemotherapy.

Exclusion Criteria:

* Contraindications to angiography and selective visceral catheterization
* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs
* Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop or mitigate such flow (ex. placing catheter distal to gastric vessels)
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Severe liver dysfunction or pulmonary insufficiency
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Pregnancy

Patients will be excluded: if they have a co-morbid disease or an acute or chronic condition that would preclude safe delivery of TheraSphere treatment and place the patient at undue risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Yung-Ho Sze, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States